Comparison of Different Techniques on First Attempt Success in Difficult Vascular Access Patients

NCT04821362

July 3, 2018

**Statistical Analyses Plan:** 

Statistical analyses will be performed using the IBM SPSS Statistics for Windows, Version 25.0. Armonk, NY: IBM Corp. The suitability of continuous variables to normal distribution will be examined using analytical methods (Kolmogorov–Smirnov). Descriptive analysis will be performed using the median and interquartile range for non-normally distributed variables and means and standard deviations for normally distributed variables. In the comparison of independent groups, Kruskal–Wallis tests will be used for non-normally distributed data. The Mann-Whitney U test will be performed to test the significance of pairwise differences for multiple comparisons using Bonferroni correction. For categorical variables, the difference between groups will be evaluated with the Chisquare test. A p-value less than 0.05 will be considered to show a statistical result.